CLINICAL TRIAL: NCT05452265
Title: Different Approach of Minimal Invasive Surgery for Gastric Subepithelial Tumor From A Single-Center Experience
Brief Title: Minimal Invasive Surgery for Gastric Subepithelial Tumor
Status: Completed | Type: Observational
Sponsor: Changhua Christian Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 220117
Record Dates: First submitted 2022-06-29; First posted 2022-07-11 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Gastric Subepithelial Tumor
Keywords: gastric subepithelial tumors; endoscopic resection; laparoscopic resection
MeSH Terms: interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- endoscopic resection (ER): ER with backup surgery was indicated for patients with endoscopic intent, and a small tumor size tolerated endoscopic retrieval.
  Interventions: Procedure: Endoscopic resection
- laparoscopic resection (LR): LR was indicated for patients with surgical intent, and those with the following conditions, which were not suitable for ER: (1) large tumor size with difficult endoscopic retrieval ; (2) symptoms of gastrointestinal tract bleeding with difficulty in endoscopic visualization; (3) suspicion of tumor rupture that required intra-abdominal exploration; and (4) histologic diagnosis of GIST with initial treatment of target therapy.

INTERVENTIONS:
Procedure: Endoscopic resection — Complete resection of gastric SETs was recommended if the tumor size was >2 cm, presence of malignant features, or if the patient was symptomatic, declined periodical surveillance, and preferred to undergo diagnostic and therapeutic resection.
  Other Names: Laparoscopic resection
  Groups: endoscopic resection (ER)

SUMMARY:
The investigators conducted a retrospective study of those patients with gastric SETs receiving ER or LR at the operative theater in the single institution from January 2013 to December 2021. Medical records were retrospectively reviewed to define patient/tumor characteristics and operative outcomes.

ELIGIBILITY:
Inclusion Criteria:

* patients with gastric subepithelial tumors
* patients received minimal invasive surgery (endoscopy or laparoscopy) for tumor resection

Exclusion Criteria:

* patients had gastric anatomic changes due to previous surgery
* patients converted open surgery

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with gastric SETs who underwent ER or LR at the operative theater in our institution
Sampling Method: Probability Sample
Enrollment: 194 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Procedure duration | during the procedure/surgery
  minutes of procedure time
Length of hospital stay | upto one month after surgery
  days of hospitalization
Rate of postoperative major complications | upto one month after surgery
  complications required further intervention, clavien dindo classification upto Grade III

IPD SHARING:
Plan to Share IPD: No